CLINICAL TRIAL: NCT03218501
Title: A Phase II, Double-Blind, Randomized, Placebo-Controlled Study of SK-1405 in Hemodialysis Patients With Uremic Pruritus
Brief Title: A Study of SK-1405 in Hemodialysis Patients With Uremic Pruritus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanwa Kagaku Kenkyusho Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MO1003
Record Dates: First submitted 2017-07-13; First posted 2017-07-14 (Actual); Last update posted 2019-03-08 (Actual); Status verified 2018-11

CONDITIONS: Uremic Pruritus in Hemodialysis Patients
Keywords: Uremic Pruritus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SK-1405 high dose (Active Comparator): SK-1405 high dose is to be administered orally once daily for 2 weeks
  Interventions: Drug: SK-1405 high dose
- SK-1405 low dose (Active Comparator): SK-1405 low dose is to be administered orally once daily for 2 weeks
  Interventions: Drug: SK-1405 low dose
- Placebo (Placebo Comparator): Placebo is to be administered orally once daily for 2 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SK-1405 high dose — SK-1405 high dose is to be administered orally once daily for 2 weeks
  Arms: SK-1405 high dose
Drug: SK-1405 low dose — SK-1405 low dose is to be administered orally once daily for 2 weeks
  Arms: SK-1405 low dose
Drug: Placebo — Placebo is to be administered orally once daily for 2 weeks
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety and dose response of SK-1405 for the treatment of subjects with uremic pruritus receiving hemodialysis, during 2 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Receiving hemodialysis three times a week for at least 12 weeks
* Worst itching VAS in a day is 30 mm or more at least 5 days during the first observation period
* Mean worst itching VAS is 50 mm or more in both the first and second observation periods

Exclusion Criteria:

* Complications that may affect the assessment of uremic pruritus
* Started or changed pruritus treatment within 13 days prior to starting observations
* Received ultraviolet treatment within 27 days prior to starting observations
* Uncontrollable hypertension, serious liver disease, serious heart disease, stroke, or malignant tumor
* Depression, schizophrenia, dementia, epilepsia, convulsive seizure, drug addiction, or alcoholism
* Pregnancy, or breastfeeding

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 269 (Actual)
Dates: Start 2017-08-28 (Actual); Primary Completion 2018-05-25 (Actual); Study Completion 2018-05-25 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Worst-itching Visual Analog Scale (VAS) | 2 weeks

SECONDARY OUTCOMES:
Change from baseline in Worst-itching Visual Analog Scale (VAS) | 1 week, 3 weeks
Change from baseline in Itch Severity Assessment | 1 week, 2 weeks, 3 weeks
Change from baseline in Sleep Quality Assessment | 1 week, 2 weeks, 3 weeks
Change from baseline in 5D Itch Scale | 2 weeks
Number of Participants with Adverse Events | 5 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Investigational site (there may be other sites in this country), Tokyo, Japan